CLINICAL TRIAL: NCT02503566
Title: Assessment of Cardiac Allograft Vasculopathy (CAV) by Optical Coherence Tomography (OCT)
Brief Title: Assessment of Cardiac Allograft Vasculopathy by Optical Coherence Tomography
Acronym: EARLY-OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institute for Clinical and Experimental Medicine (Other Government)
Collaborators: St. Anne (Unknown)
Responsible Party: Principal Investigator, Michal Pazdernik, MD, M.D., Institute for Clinical and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KKIKEM
Record Dates: First submitted 2015-07-15; First posted 2015-07-21 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Disorder Related to Cardiac Transplantation
Keywords: CAV; OCT; heart rate; antibodies
MeSH Terms: interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): Optical coherence tomography will be performed in all patients
  Interventions: Device: Optical coherence tomography

INTERVENTIONS:
Device: Optical coherence tomography — Optical coherence tomography performed during regular coronary angiography

SUMMARY:
Cardiac allograft vasculopathy (CAV) is characterized by marked intimal proliferation and concentric vascular thickening and fibrosis. CAV remains the leading cause of late morbidity and mortality in heart transplant recipients. Optical coherence tomography (OCT) is a new generation catheter-based modality that acquires images at a spatial resolution of 10-20 μm which is 10-fold greater than that of intravascular ultrasound (IVUS). OCT is currently the most sensitive imaging technique for early CAV detection. Recent studies proved that circulating human leukocyte antigen (HLA) directed donor-specific antibodies correlate with increased mortality and CAV. Contradiction of scientific results has been reported regarding increased resting heart rate and development of CAV. Larger prospective studies using more sensitive CAV detecting methods are required to enhance our understanding. Novel immunosuppressants, mechanistic target of rapamycin (mTOR) inhibitors, may attenuate CAV progression and may improve long-term allograft survival owing to favorable coronary remodeling.

Aim of the study: Use OCT imaging for identification of patients with early rapid progression of CAV (rapid progressors) and to identify the critical risk factors responsible for CAV progression. The impact of conventional and heart transplant (HTx) specific risk factors, such as donor-specific antibodies or rapid heart rate will be studied in a prospective, national-level cohort study. The implication of OCT results will lead to adjustment of immunosuppressive therapy in one year after heart transplant to prevent further progression of the disease in CAV rapid progressors.

Working hypotheses:

1. Patients with rapid progression of cardiac allograft vasculopathy can be identified by increased titers of donor specific anti-human leukocyte antigen (anti-HLA) and/or antibodies against major histocompatibility complex (MHC) class I-related chain A (MICA) antibodies.
2. Specific high-risk characteristics of anti-HLA antibodies can be identified that are associated with particularly high rate of CAV progression (vascular complement activation in biopsies, certain HLA haplotypes).
3. Tachycardia in heart transplant recipients represents a risk factor for development of cardiac allograft vasculopathy.
4. Influence of anti-HLA antibodies and increased heart rate is independent of already established risk factors of CAV.

DETAILED DESCRIPTION:
Cardiac allograft vasculopathy (CAV) represents the leading cause of late morbidity and mortality in heart transplant recipients and accounts for a second of all-cause mortality at 3 years. Development of CAV is a complex process involving intimal thickening, atherosclerosis, thrombosis and vasculitis by histology, but ultimately, intimal hyperplasia is the predominant cause of lumen narrowing, leading to ischemia and graft failure. In distinction from general coronary atherosclerosis, which is marked by focal and eccentric fibrofatty atheroma, CAV affects diffusely the entire coronary vasculature with marked intimal proliferation and concentric vascular thickening and fibrosis.

Optical coherence tomography (OCT), compared with IVUS, is more sensitive for early detection of CAV. OCT is a new generation catheter-based modality that acquires images at a spatial resolution of 10-20 μm which is 10-fold greater than that of IVUS. OCT could obviously identify the layer of media as a lower-echoic line, which could not be identified by IVUS. When assessing the quality of an intracoronary structure accurately, OCT seems to have more potential than IVUS.

The endothelial cells of the cardiac vasculature express human leukocyte antigens (HLA) and others, such as vimentin and major histocompatibility complex (MHC) class I-related chain A (MICA), and appear to be primary targets of cell-mediated and humoral immune responses after heart transplant (HTx). Circulating antibodies mediate rejection through complement activation and fixation on graft endothelium, thereby predisposing the patient to graft loss, accelerated cardiac allograft vasculopathy, and death. The rate of allosensitized patients (patients with circulating antibodies against donor antigens) on waiting lists is increasing as a consequence of growing numbers of retransplants and assist-device implantations. Allosensitization is a consequence of exposure to disparate HLA molecules during pregnancy, blood/platelet transfusions, or after cardiac repairs with homograft material, but may occur in some patients even without any of these triggers from unknown reasons.

Orthotopic heart transplantation is accompanied by sympathetic and parasympathetic denervation. The subsequent heart rate is usually higher and the circadian variation is low due to elimination of the vagus nerve effect. It is known that persistent increase in heart rate contributes to the pathogenesis of vascular diseases.

AIMS OF THE PROJECT The aim of this study is to use OCT imaging for identification of patients with early rapid progression of cardiac allograft vasculopathy (rapid progressors) and to identify the critical risk factors responsible for CAV progression. The impact of conventional and HTx-specific risk factors, such as donor-specific antibodies (using the most sensitive methods for its measurement) or rapid heart rate (using repeated Holter monitoring) will be studied in a prospective, national-level cohort study. The implication of OCT results will lead to adjustment of immunosuppressive therapy in one year after heart transplant to prevent further progression of the disease in CAV rapid progressors.

WORKING HYPOTHESES

1. Patients with rapid progression of cardiac allograft vasculopathy can be identified by increased titers of donor specific anti-HLA and/or MICA antibodies.
2. Specific high-risk characteristics of anti-HLA antibodies can be identified that are associated with particularly high rate of CAV progression (vascular complement activation in biopsies, certain HLA haplotypes).
3. Tachycardia in heart transplant recipients represents a risk factor for development of cardiac allograft vasculopathy.
4. Influence of anti-HLA antibodies and increased heart rate is independent of already established risk factors of CAV.

STUDY DESIGN Collection of data and blood samples will be performed at the same time as the patient's regularly scheduled surveillance cardiac catheterization (1 month and 12 months after heart transplant). Additionally donor-specific anti-HLA antibodies (class I, II) and MHC complex class I - related chain A (MICA) antibodies will be measured also before heart transplant and in 6 months after heart transplant during regular follow-ups.

OCT (optical coherency tomography) imaging will be performed at the same time as the patient's regularly scheduled surveillance cardiac catheterization (1 month and 12 months after heart transplant). OCT imaging will be performed with the commercially available second-generation frequency domain Ilumien Optis (St. Jude Medical, St. Paul, MN). The OCT catheter (Dragonfly Duo) will be advanced over a 0.014-inch coronary guide wire into the middle segments of all three main arteries (left anterior descending, left circumflex and right coronary artery) and imaging will be performed by automated pullback with a length 45 mm, with pullback speed 25 mm/sec in high resolution mode (10 frames /mm). OCT examination will be performed after administration of 200-300 μg of intracoronary nitroglycerin and simultaneous injection of 14 ml of contrast agent to each artery by power injector through the guiding catheter. OCT data will be used for 3-D vessel reconstruction done by the fusion with routine angiography performed in two projections at least 60 degree apart.

The image data acquired from two-plane angiography, can be utilized to accurately reconstruct the path and orientation of the OCT catheter in 3-D.

The two-plane angiograms are taken immediately prior to the pullback start and cover at least one heart cycle each. They are used to extract the catheter path automatically along the expected pullback trajectory by a dynamic programming approach. From the known imaging geometry, an accurate 3-D model of the catheter path within the respective vessel segment is generated for end-diastolic heart phase. For OCT acquisition, motorized pullback ensures a constant pullback speed, thus allowing to assign each OCT image frame a specific location on the 3-D catheter trajectory model. The relative and absolute orientations of the OCT frames are determined using previously reported system for establishing the absolute orientation in 3-D on IVUS images. Quantitative data can be derived from the contour data, such as luminal dimensions and plaque-cap thickness, actually considering the vessel curvature in contrast to conventional OCT reconstruction systems. The space between adjacent contours is interpolated to form a volume element. In locations of the plaque cap, integrating over an entire vessel segment or any part thereof yields the total plaque cap volume enclosed by the inner and outer cap surfaces.

The OCT examination will be analyzed according to OCT consensus standard definitions. Intima can be recognized as a uniform signal-rich bright layer and media as a signal-poor darker layer due to low backscatter. The lumen, intima, and media layers will be traced automatically with manual correction to obtain average thickness and areas for every frames. The only segment without any signs of coronary atherosclerosis on coronary angiography will be used for OCT examination. Following indices will be analyzed:

1. Normalized intimal volume: the sum of intimal cross sectional area (difference between media area and lumen area) in every frames / pullback length.
2. Normalized lumen volume: the sum of lumen cross sectional area in every frames / pullback length.
3. Mean intima thickness: the values from all sufficient quality frames will be averaged to yield average intima thickness.
4. Mean intima-to-media ratio (I/M): Values from all sufficient quality frames will be averaged to yield average intima thickness, and media thickness. The intima-to-media ratio (I/M) will be calculated as a ratio of average area of each layer over the whole pullback. An I/M ratio of more than 1 will be defined as abnormal.

These indices will be compared between baseline and follow-up examinations. After identification of vascular landmarks corresponding in the two 3-D vessel models, the patient specific model pairs will be co-registered to correctly match the OCT pullbacks.

OCT baseline and follow-up examinations will be performed in Prague (IKEM hospital) and Brno (Saint Anna hospital) and data will be send to the core lab in the Iowa Institute for Biomedical Imaging, The University of Iowa, USA for analysis. Iowa Institute for Biomedical Imaging is a research centre, which has extensive experience with the evaluation of coronary atherosclerosis. For the purpose of detailed analysis of the coronary arteries unique software for creating 3-D reconstructions of coronary arteries based on the fusion of angiography and optical coherence tomography was developed at this institution. This software enables exact assessment of plaque and lumen volumes. Software is protected by U.S. patent. Because of large volume of data and patients in this project, applications of such automated analytic tools are prerequisite of successful accomplishment.

Mean heart rate will be measured during 24 hour ECG Holter monitoring, which will evaluate all necessary parameters including its circadian variability. ECG Holter recordings will be performed in 1 month and in 12 months after heart transplant. In addition to mean 24 hour heart rate, time and frequency domain components of heart rate variability will be analyzed to obtain estimate the extent of vagal reinnervation.

Donor-specific anti-HLA antibodies(class I,II) and MHC complex class I - related chain A (MICA) antibodies will be measured (before heart transplant, 1 month, 6 months and 12 months after heart transplant). Evaluation of anti-HLA antibodies levels (titers) in the serum of a patient is performed by fluorescence intensity of formed complexes. Double laser cytometer Luminex 100 IS 2.3 is used for fluorescence reading. Based on comparison of negative and positive controls, cut-off is calculated.

Conventional risk factors for CAV will be determined in 1 month and in 12 months after heart transplant.

Lipid profile (total cholesterol, LDL, HDL and triglycerides) will be measured. Blood pressure in triplicate will be measured in supine position (1 hour before regular endomyocardial biopsies). Glycemic control will be quantified by measurements of Hemoglobin A1 level, plasma glucose. Cytomegalovirus (CMV) status will be measured by immunoglobulin G (IgG), immunoglobulin M (IgM) titers.

Other monitored parameters will be: 1) the post transplant course and clinical status; the occurrence of graft dysfunction (echocardiographic monitoring will follow each endomyocardial biopsy), 2) the occurrence of cellular and/or humoral rejection in endomyocardial biopsies (8 protocolar endomyocardial biopsies within 12 months after heart transplantation), 3) presence and tissue distribution (vascular/non-vascular) staining for complement fragments C3 and C4 (markers of antibodies-mediated complement activation), 4) the period of cardiac allograft cold ischemia 5) aetiology of brain death of the donor 6) degree of HLA mismatch between donor and recipient, 7) blood cytokine levels involved in regulation of humoral immune response.

ELIGIBILITY:
Inclusion Criteria:

* All new cardiac transplant recipients ≥18 years

Exclusion Criteria:

* Severe renal dysfunction (GFR less than 30 ml/min)
* Active infection
* Active cellular/humoral rejection
* Unwilling or unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09-01 (Actual); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Rapid progression of cardiac allograft vasculopathy | 1 year
  OCT imaging will be used for identification of patients with early rapid progression of cardiac allograft vasculopathy. Normalized intimal volume, normalized lumen volume, mean intima thickness and mean intima-to-media ratio (I/M) will be used to identify fast progression of CAV.

SECONDARY OUTCOMES:
Donor specific anti-HLA and/or MICA antibodies | 1 year
  Patients with rapid progression of cardiac allograft vasculopathy can be identified by increased titers of donor specific anti-HLA and/or MICA antibodies. Evaluation of anti-HLA antibodies levels (titers) in the serum of a patient is performed by fluorescence intensity of formed complexes. Double laser cytometer Luminex 100 IS 2.3 is used for fluorescence reading.
Heart rate | 1 year
  Tachycardia in heart transplant recipients might represents a risk factor for development of cardiac allograft vasculopathy. Mean heart rate will be measured during 24 hour ECG Holter monitoring, which will evaluate all necessary parameters including its circadian variability.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Pazdernik, M.D., Principal Investigator — Institute for Clinical and Experimental Medicine
Locations (2):
- Czechia (2):
  - Helena Bedanova, Brno
  - Michal Pazdernik, Prague

REFERENCES:
- [Background] Costanzo MR, Naftel DC, Pritzker MR, Heilman JK 3rd, Boehmer JP, Brozena SC, Dec GW, Ventura HO, Kirklin JK, Bourge RC, Miller LW. Heart transplant coronary artery disease detected by coronary angiography: a multiinstitutional study of preoperative donor and recipient risk factors. Cardiac Transplant Research Database. J Heart Lung Transplant. 1998 Aug;17(8):744-53. PMID 9730422
- [Background] Stehlik J, Edwards LB, Kucheryavaya AY, Aurora P, Christie JD, Kirk R, Dobbels F, Rahmel AO, Hertz MI. The Registry of the International Society for Heart and Lung Transplantation: twenty-seventh official adult heart transplant report--2010. J Heart Lung Transplant. 2010 Oct;29(10):1089-103. doi: 10.1016/j.healun.2010.08.007. No abstract available. PMID 20870164
- [Background] Wehner J, Morrell CN, Reynolds T, Rodriguez ER, Baldwin WM 3rd. Antibody and complement in transplant vasculopathy. Circ Res. 2007 Feb 2;100(2):191-203. doi: 10.1161/01.RES.0000255032.33661.88. PMID 17272820
- [Background] Kaczmarek I, Deutsch MA, Kauke T, Beiras-Fernandez A, Schmoeckel M, Vicol C, Sodian R, Reichart B, Spannagl M, Ueberfuhr P. Donor-specific HLA alloantibodies: long-term impact on cardiac allograft vasculopathy and mortality after heart transplant. Exp Clin Transplant. 2008 Sep;6(3):229-35. PMID 18954302
- [Background] Palatini P, Julius S. Elevated heart rate: a major risk factor for cardiovascular disease. Clin Exp Hypertens. 2004 Oct-Nov;26(7-8):637-44. doi: 10.1081/ceh-200031959. PMID 15702618
- [Background] Olmetti F, Pinna GD, Maestri R, D'Armini A, Pellegrini C, Vigano M, Lilleri D, Gerna G, Febo O, La Rovere MT. Heart rate and cardiac allograft vasculopathy in heart transplant recipients. J Heart Lung Transplant. 2011 Dec;30(12):1368-73. doi: 10.1016/j.healun.2011.07.009. Epub 2011 Aug 15. PMID 21840733
- [Background] Keogh A, Richardson M, Ruygrok P, Spratt P, Galbraith A, O'Driscoll G, Macdonald P, Esmore D, Muller D, Faddy S. Sirolimus in de novo heart transplant recipients reduces acute rejection and prevents coronary artery disease at 2 years: a randomized clinical trial. Circulation. 2004 Oct 26;110(17):2694-700. doi: 10.1161/01.CIR.0000136812.90177.94. Epub 2004 Jul 19. PMID 15262845
- [Background] Garrido IP, Garcia-Lara J, Pinar E, Pastor-Perez F, Sanchez-Mas J, Valdes-Chavarri M, Pascual-Figal DA. Optical coherence tomography and highly sensitivity troponin T for evaluating cardiac allograft vasculopathy. Am J Cardiol. 2012 Sep 1;110(5):655-61. doi: 10.1016/j.amjcard.2012.04.047. Epub 2012 May 26. PMID 22640973